CLINICAL TRIAL: NCT00918697
Title: Mechanical Versus Alcohol-Assisted Epithelial Debridement During Photorefractive Keratectomy: A Confocal Microscopic Clinical Trial
Brief Title: Mechanical Versus Alcohol Epithelial Debridement During Hotorefractive Keratectomy (PRK)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Ophthalmic Research Center,, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 8713
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-04

CONDITIONS: Refractive Error; Myopia
Keywords: photorefractive keratectomy; PRK; alcohol-assisted debridement; mechanical debridement; confocal scan; confocal microscopy
MeSH Terms: conditions — Refractive Errors; Myopia | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Mechanical debridment (Active Comparator): In this arm, corneal epithelium was removed during PRK using conventional mechanical method.
  Interventions: Procedure: Mechanical debridement
- Alcohol-asstisted debridement (Experimental): In this arm, corneal epithelium was removed using ethanol 20% during PRK.
  Interventions: Procedure: Alcohol-assisted debridement

INTERVENTIONS:
Procedure: Mechanical debridement — For mechanical epithelial removal, an 8.0-mm optical zone marker was applied to the cornea, centering over the entrance pupil. A hockey spatula was used to remove the central corneal epithelium.
  Arms: Mechanical debridment
Procedure: Alcohol-assisted debridement — For alcohol-assisted debridement, 20% ethyl-alcohol solution was instilled into an 8.0-mm well and kept in contact with epithelium for 20 seconds (being careful to avoid spillage over the areas not being treated). It then absorbed using a dry cellulose sponge followed by copious irrigation with BSS. The epithelium of the central cornea was removed using a blunt spatula.
  Arms: Alcohol-asstisted debridement

SUMMARY:
In this prospective randomized clinical trial, confocal microscopy was used to evaluate the effect of mechanical versus alcohol-assisted epithelial debridement during photorefractive keratectomy (PRK)on corneal cellular elements. Sixty-six eyes of 33 subjects with a spherical equivalent less than -4.00 D who completed all follow-up visits were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* spherical equivalent ≤ -4.0 D
* cylinder ≤ 1.50 D

Exclusion Criteria:

* history of ocular trauma or surgery
* any corneal and ocular pathologies
* central corneal thickness < 500 µm
* scotopic pupil diameter > 6.0 mm
* any abnormalities in corneal plain or elevation topographies favoring keratoconus or other ectatic disorders
* the presence of systemic disorders such as collagen vascular diseases

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-07; Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Corneal cellular elements.
  Confocal microscopic findings of corneal cellular elements.

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran